CLINICAL TRIAL: NCT02353936
Title: A Phase II Trial of Afatinib in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of Esophagus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0432
Record Dates: First submitted 2015-01-23; First posted 2015-02-03 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Squamous Cell Carcinoma of Esophagus
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- afatinib group (Experimental)
  Interventions: Drug: BIBW2992

INTERVENTIONS:
Drug: BIBW2992 — International Nonproprietary Name (INN): BIBW 2992 Pharmacological dosage form: Film-coated tablet Supplier: Boehringer Ingelheim Pharma GmbH & Co. KG Unit content: 40 mg, 30 mg, 20 mg film-coated tablet (BIBW 2992 content in film-coated tablet is related with equivalent free base BIBW 2992.) Daily dose: 40 mg Dosing period: To be successively administered once daily until a disease will develop, an unacceptable adverse event will occur, or another reason requiring discontinuation of the study will occur; For administration, study treatment consists of periods(each 4 weeks(28 days)).
  Route of administration: Orally (Take by swallowing) Dosage: Once daily

SUMMARY:
As a 2nd generation EGFR-TKI that irreversibly binds to EGFR receptors, afatinib showed the possibility of superior effects to 1st generation TKIs such as erlotinib and gefitinib. In a phase III study LUX-lung 3 in patients with EGFR mutation-positive non-small-cell lung cancer, afatinib monotherapy showed longer progression-free disease survival time of 11.1 months than that (6.9 months) of pemetrexed/cisplatin combination therapy. Based on such the results, it is currently recommended as the standard first-line treatment for EGFR mutation-positive lung cancer, and clinical studies are also being actively conducted in other types of carcinomas characterized by EGFR gene mutation and overexpression. Thirty (30) solid cancer patients were included in a phase I trial of afatinib, and of them, a patient with esophageal cancer had partial response. Taken together, based upon the results from clinical trials of afatinib conducted so far, 7 out of 15 esophageal cancer patients achieved clinical responses of 3 months or longer.

Hence, the overall results from previous studies of gefitinib and erlotinib as EGFR TKIs and our study of dacomitinib, as well as from preceding studies of afatinib - a 2nd generation EGFR TKI - suggest the possibility of an effective therapy in esophageal cancer characterized by well-known EGFR overexpression. In this phase II trial, afatinib shall be administered to patients with squamous cell carcinoma of esophagus to evaluate its effects and toxicity. Also, biomarkers to predict responses to afatinib shall be explored through further studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of esophagus
* Age ≥ 20
* ECOG PS 0-2
* Ineligibility for local therapy (surgery or radiotherapy)
* Patients who have failed to respond to or receive a first-line, palliative platinum-based chemotherapy

  1. Allowed to enroll the patients who have developed the recurrent cancer within 6 months after definitive/neo-adjuvant/adjuvant platinum-based chemotherapy(± radiotherapy), by considering the prior therapy as first-line chemotherapy.
  2. Allowed to enroll the patients who cannot undergo platinum-based chemotherapy or concurrent chemo-radiotherapy due to concern for renal function deterioration and the patient intolerance, without prior chemotherapy history.
* At least one bidimensionally measurable disease as defined by RECIST ver 1.1
* Adequate organ function for treatment

  1. Absolute neutrophil count (ANC) >=1000 cells/mm3
  2. Platelets ≥ 100,000 cells/mm3
  3. Estimated creatinine clearance ≥50 mL/min, or serum creatinine <1.5 x institution upper limit of normal (ULN) using Cockcroft and Gault formulas
  4. Bilirubin ≤1.5 x ULN
  5. AST (SGOT) ≤2.5 x ULN (5.0 x ULN if hepatic metastases)
  6. ALT (SGPT) ≤2.5 x ULN (5.0 x ULN if hepatic metastases)
  7. 12-Lead electrocardiogram (ECG) with normal tracing or nonclinically significant changes that do not require medical intervention QTc interval ≤470 msec and without history of Torsades de Pointes or other symptomatic QTc abnormality
* The patient who has signed the informed consent prior to conducting study related screening procedures, and who understands that the study may be discontinued at anytime without disadvantages

Exclusion Criteria:

* Previous treatment with EGFR tyrosine kinase inhibitors
* Chemotherapy , immunotherapy or investigational durg within 3 weeks of study entry
* Any major operation or irradiation within 4 weeks of baseline disease assessment
* Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug
* Patients who confirmed CNS metastasis must have completed any prior treatment for CNS metastasis and steroid therapy for brain metastasis should stopped more 1week and stabled before first dose of study treatment
* Patients with known interstitial lung disease
* Patients with uncontrolled or significant cardiovascular disease
* Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, thyroid cancer, or other solid tumors treated curatively and without evidence of recurrence for at least 3 years prior to study entry.
* Pregnant or breast feeding women
* Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
response rate | every 8 weeks until 2 years

SECONDARY OUTCOMES:
Progression free survival | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea